CLINICAL TRIAL: NCT02542501
Title: A Prospective Post Marketing Non Interventional Study to Evaluate the Presence of Lower Urinary Tract Symptoms (LUTS) in Prostate Cancer Patients Scheduled to Receive LHRH Analogues and to Evaluate the Effect of LHRH Analogues on Lower Urinary Tract Symptoms (ANALUTS Study)
Brief Title: Study to Evaluate the Presence of Lower Urinary Tract Symptoms (LUTS) in Prostate Cancer Patients Scheduled to Receive Luteinizing Hormone Releasing Hormone (LHRH) Analogues
Acronym: ANALUTS
Status: Completed | Type: Observational
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: A-ES-52014-219
Record Dates: First submitted 2015-07-07; First posted 2015-09-07 (Estimated); Last update posted 2018-12-21 (Actual); Status verified 2018-12

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The intention of this study is to investigate how many patients with prostate cancer, planned to be treated with LHRH analogues without history of surgery or radiotherapy, are suffering from LUTS. In addition the effect of LHRH analogues on the improvement of theses primary LUTS symptoms over time will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Adult men with locally advanced or metastatic prostate cancer scheduled to receive LHRH analogues. A patient who has completed an IPSS questionnaire in his last visit, before the start of LHRH analogues, will be able to participate in the study. This last visit has to be done 6 months before the baseline visit.
* Patients having provided written informed consent
* Patients mentally fit for completing a self-administered questionnaire

Exclusion Criteria:

* Any surgical or radiotherapy treatment performed at prostate level before the entry of the study
* Patient with castrate levels of testosterone ( < 50 ng/dL) at his first IPSS questionnaire
* Patients who are also participating in any other clinical study within the last 2 months before study entry
* Life expectancy of less than 12 months

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 470 (Actual)
Dates: Start 2015-07; Primary Completion 2018-07-21 (Actual); Study Completion 2018-07-21 (Actual)

PRIMARY OUTCOMES:
The number of patients having Lower Urinary Tract Symptoms (LUTS) at baseline. | Baseline
The percentage of patients suffering from prostate cancer with moderate to severe LUTS (International prostate symptom score (IPSS) >7) at baseline and having at least 3 points reduction of IPSS score at the end of study (48 weeks). | Week 48

SECONDARY OUTCOMES:
The percentage of patients suffering from prostate cancer with moderate to severe LUTS (score IPSS > 7) at baseline and having at least 3 points reduction of IPSS score at week 24. | Week 24
The correlation between IPSS score changes and total prostatic-specific antigen (PSA) changes after 24 weeks of treatment compared to baseline in patients with non-operable prostate cancer presenting moderate to severe LUTS (score IPSS >7) at baseline. | Week 24
  Assessed with the Pearson correlation coefficient
The correlation between IPSS score changes and total PSA changes after 48 weeks of treatment compared to baseline in patients with non-operable prostate cancer presenting moderate to severe LUTS (score IPSS >7). | Week 48
  Assessed with the Pearson correlation coefficient
Comparison of the percentage of patients presenting an IPSS ≥ 3 at week 24 to the percentage of patients presenting an IPSS ≥ 3 at baseline. | Week 24
  Assessed with the McNemar's test
Comparison of the percentage of patients presenting an IPSS ≥ 3 at week 48 to the percentage of patients presenting an IPSS ≥ 3 at baseline. | Week 48
  Assessed with the McNemar's test

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (32):
- Portugal (5):
  - Hospital Universitário de Coimbra, Coimbra
  - Hospital de São José, Lisbon
  - Hospital de Santa Maria, Lisbon
  - Hospital Pedro Hispano, Matosinhos Municipality
  - Hospital Geral de Santo António, Porto
- Spain (27):
  - Hospital Esperit Sant, Santa Coloma de Gramenet, Barcelona
  - Hospital Sureste, Arganda, Madrid
  - Hospital Universitario A Coruña, A Coruña
  - Hospital Germans Trias I Pujol, Badalona
  - H. del Mar, Barcelona
  - H. Valle Hebrón, Barcelona
  - Hospital de Basurto, Bilbao
  - Hospital de Ciudad Real, Ciudad Real
  - Hospital Getafe, Getafe
  - H. Bellvitge, L'Hospitalet de Llobregat
  - Hospital de León, León
  - Hospital de la Princesa, Madrid
  - Hospital Univ. La Paz, Madrid
  - Hospital del Sureste, Arganda de Rey, Madrid
  - Hospital Althaia, Manresa
  - H. Parc Tauli, Sabadell
  - Hospital de Salamanca, Salamanca
  - Hospital de Donosti, San Sebastián
  - Hospital Infanta Sofía, San Sebastián de los Reyes
  - H. Univ. Nuestra Señora de la Candelaria, Santa Cruz de Tenerife
  - Complejo Clínico Universitario de Santiago, Santiago de Compostela
  - Hospital Joan XXIII, Tarragona
  - Hospital Clínico de Valladolid, Valladolid
  - Hospital Universitari de Vic, Vic
  - H. Do Meixoeiro, Vigo
  - Hospital Santiago Apóstol, Vitoria-Gasteiz
  - Hospital de Txagorritxu, Vitoria-Gasteiz